CLINICAL TRIAL: NCT00612443
Title: Healing Touch and Health-Related Quality of Life in Women With Breast Cancer in Women With Breast Cancer Receiving Radiation Therapy
Brief Title: Healing Touch and Health-Related Quality of Life in Women With Breast Cancer Receiving Radiation Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Lisa L Schnepper MSN, FNP-BC PhD candidate, University of Wisconsin-Milwaukee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07.0.243; 07-006400
Record Dates: First submitted 2008-01-25; First posted 2008-02-11 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Breast Neoplasms
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Touch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): non-contact Healing Touch treatment for 20-30 minutes once a week during the course of radiation therapy
  Interventions: Behavioral: Healing Touch
- 2 (Sham Comparator): A RN graduate assistant will provide a sham treatment of 20-30 minutes of presence.
  Interventions: Behavioral: Sham treatment

INTERVENTIONS:
Behavioral: Sham treatment — The sham/placebo treatment will consist of the RN graduate assistant standing near the table, slowly walking around from each side and to the foot of the table stopping periodically. The RN graduate assistant will be instructed to not focus on the patient in thought. While providing the placebo treatment the RN graduate assistant will mentally do multiplication equations. This serves as a distracter to keep the RN graduate assistant from setting intention or thoughts on the participant. At no time will the RN performing the placebo treatment move hands or arms over or around the participant or come in physical contact with the participant. The placebo treatment will be a minimum of 20 minutes but no greater than 30 minutes in length. A timer will be set in the treatment room to notify the practitioner of the time limit.
  Other Names: placebo treatment
  Arms: 2
Behavioral: Healing Touch — Behavioral: Healing Touch The Healing Touch intervention will consist of a brief meditative state in which the practitioners sets the intention of healing for the session. A hand scan to assess the biofield; consists of a technique of where the practitioner slowly moves her hands three to six inches above the body going from head to toe, to assess for any disturbances in the biofield; a non-contact Healing Touch treatment which will follow, to include a connection of the chakras. The chakras are connected by placing the hands above the body over each chakra, starting at the feet and progressing to the head. This will be followed by smoothing the biofield, achieved by the Practitioner slowly moving her hands above the body from the head and moving towards the feet (Hover-Kramer et al., 1996). At no time will the Practitioner make physical contact with the participant during the treatment. The treatment will be 20 minutes to 30 minutes in length.
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Healing Touch to improve health-related quality of life in women with breast cancer receiving radiation therapy.

Research Hypothesis Healing Touch significantly improves health-related quality of life when compared to a placebo treatment, among women receiving radiation therapy for treatment of breast cancer.

DETAILED DESCRIPTION:
Purpose/objective The purpose of this study is to evaluate the efficacy of the CAM biofield therapy of Healing Touch to improve health-related quality of life (HRQOL) in women with breast cancer receiving radiation therapy. The proposed study will build on existing research by Cook, Guerrio and Slater (2004) who studied Healing Touch and HRQOL in women receiving radiation therapy for breast and gynecologic cancers. Outcome measures of HRQOL as measured by Short Form-36 (SF-36) tool were used (Norris et al. 2004). The SF-36 is a tool to measure HRQOL, a 36 item tool that measures nine domains of health: a) functional limitations in physical activity secondary to health problems, b) limitations in social activity secondary to physical or mental health issues, c) limitation in role activities secondary to physical health problems, d) limitation in role activities secondary emotional health problems, e) to pain, f) overall mental health, g) vitality, h) perceptions of health and i) health transitions (Norris et. al., 2004). Measurements were taken at baseline and end of study.

Cook et al (2004) found that all women in the study had improved scores on the HRQOL Short Form-36 (SF-36) tool used (Norris et al. 2004). Equally important, the women who received Healing Touch had greater improvement in all subscale scores in comparison to placebo treatment. The overall score on the SF-36 (p value .00) and areas of emotional role functioning (p value .00), mental health (p value .03) and health transitions (p value .00) had statistical significance in the Healing Touch treatment group. The placebo treatment group had statistical significance in the areas of physical role functioning (p value .00) and health transition (p value .01).In group comparisons of mean SF-36 scores, the Healing Touch group had statistically greater improvement, than the placebo group, with a p value of < .05, in the areas of physical functioning, pain and vitality.

The total number of participants in the study was 62 women, with 38 who had gynecologic cancers and 24 participants with breast cancer. The number of breast cancer patients was inadequate to perform a separate statistical analysis of this sub-group (Cook et al., 2004). Therefore, this study will specifically focus on women with breast cancer to investigate the efficacy of using Healing Touch to improve HRQOL improvement in women with breast cancer receiving radiation therapy.

Research Aims The research aim of the proposed study is to determine the efficacy of Healing Touch in significantly improving HRQOL, as measured by the Functional Assessment of Cancer Therapy-Breast (FACT-B)(Brady et al., 1997; Cella et al., 1993) scale among women receiving radiation therapy for breast cancer treatment (see Appendix A for FACT-B; see Appendix B for FACT-B scoring).

Research Hypothesis Healing Touch significantly improves HRQOL, as measured by the FACT-B, when compared to a placebo treatment, among women receiving radiation therapy for treatment of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Any female patient being treated with radiation therapy for a diagnosis of stage 0, I, or II breast cancer
* Aged 18 years or greater
* Understands written and spoken English
* receiving 4, 5 or 6 weeks of radiation are eligible with a minimum study enrollment time of 4 weeks.

Exclusion Criteria:

* Anyone not meeting the above

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the difference in the FACT-B total score from baseline, midpoint and end of study participation. | Measurement at study entrance, after 3 weeks and study exit (4, 5 or 6 weeks).

SECONDARY OUTCOMES:
Secondary endpoints are the sub-scales of the FACT-B scores physical well- being, social/family well-being, emotional well-being, functional well-being,and breast cancer subscales) | study entrance, after 3 weeks and at study exit

CONTACTS AND LOCATIONS:
Overall Officials: Lisa L Schnepper, MSN, PhD (c), Principal Investigator — University of Wisconsin, Milwaukee; Laura M Anderko, PhD, Study Chair — University of Wisconsin, Milwaukee
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States